CLINICAL TRIAL: NCT07098078
Title: Domperidone Dose and the Risk of Serious Adverse Events in Older Adults With Advanced Chronic Kidney Disease: A Population-Based Cohort Study Research Protocol
Brief Title: Domperidone and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 594 000; ICES # 2025 0906 594 000 (Other: Canadian Institutes of Health Research)
Record Dates: First submitted 2025-06-06; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: chronic kidney disease; high-throughput computing; domperidone; adverse events; older adults
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Domperidone; Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low dose of domperidone <30 mg/day: Residents of Ontario and Alberta aged 66 years or older with advanced CKD with an eGFR of less than 45 mL/min/1.73m² (excluding individuals undergoing dialysis or those who have received a kidney transplant) who have filled a new oral prescription for domperidone (low dose <30mg/day) at an outpatient pharmacy under Ontario Drug Benefit (ODB) program from January 1, 2008, to September 30, 2024. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once. The accrual period for Alberta will be determined.
  Interventions: Drug: Domperidone (drug)
- High dose of domperidone ≥ 30 mg/day: Residents of Ontario and Alberta aged 66 years or older with advanced CKD with an eGFR of less than 45 mL/min/1.73m² (excluding individuals undergoing dialysis or those who have received a kidney transplant) who have filled a new oral prescription for domperidone (high dose ≥ 30 mg/day) at an outpatient pharmacy under Ontario Drug Benefit (ODB) program from January 1, 2008, to September 30, 2024. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once. The accrual period for Alberta will be determined.
  Interventions: Drug: Domperidone (drug)

INTERVENTIONS:
Drug: Domperidone (drug) — The primary exposure of interest will be oral domperidone at a dose of 30 mg or more per day, which represents the median dose found in high-throughput computing analyses. For the primary comparison, oral domperidone at doses below 30 mg per day will be chosen to reduce the influence of indication bias.
  Other Names: APO-Domperidone; BIO-Domperidone; Domperidone-10; GMD-Domperidone; JAMP-Domperidone; Mar-Domperidone; PMS-Domperidone [DSC]; Priva-Domperidone [DSC]; PRZ-Domperidone; TARO-Domperidone; TEVA-Domperidone

SUMMARY:
This study will assess whether initiating domperidone at doses ≥30 mg/day compared to <30 mg/day in patients with advanced chronic kidney disease (CKD) (estimated glomerular filtration rate [eGFR] <45 mL/min/1.73 m² but not receiving dialysis) is associated with a higher 30-day risk of a composite outcome of all-cause hospitalization or all-cause emergency visits or all-cause mortality.

DETAILED DESCRIPTION:
*Summary*

Background: Domperidone is a dopamine antagonist used to relieve symptoms of upper gastrointestinal motility disorders, such as nausea, vomiting, and delayed gastric emptying. Its use in patients with chronic kidney disease (CKD) may increase the risk of adverse events. However, current prescribing guidelines and product monographs provide conflicting recommendations for dosing in this at-risk population, leading to uncertainty about the appropriate use of domperidone in patients with CKD. The investigators have recently developed a novel high-throughput computing approach to identify medications that may harm patients with CKD using healthcare databases from Ontario. High-throughput study findings suggest that older adults who are newly prescribed domperidone face an increased risk of adverse outcomes compared to a similar cohort of non-users. To confirm these signals, the investigators will conduct a population-based cohort study among older adults with advanced CKD across two Canadian provinces: Ontario and Alberta.

Methods: The investigators will conduct a retrospective cohort study using large provincial administrative healthcare databases from Ontario and Alberta, Canada. The study will include older adults (≥66 years of age) who received a prescription for oral domperidone between 2008 and 2024. In Ontario, the sample will be accrued from January 1, 2008, through September 30, 2024. In Alberta, the accrual period will be determined based on data availability. The prescription date will be the index date (start of cohort follow-up). Patients with CKD initiating treatment with domperidone will be divided into two groups based on their dosage: high dose (≥ 30 mg/day) and low dose (<30 mg/day). The investigators will use propensity score weighting to ensure groups are comparable across baseline characteristics. Patient outcomes will be assessed 30 days following the index date. Modified Poisson regression will be used to compute the risk ratio (95% Confidence interval (CI)), and binomial regression will be used to compute the risk difference (95% CI) using the weighted cohort, with the low-dose group as the referent.

*Literature Review*

Domperidone, a peripheral dopamine-2 receptor antagonist with gastrokinetic and antiemetic effects, was first marketed in Canada in 1985 as Motilium, which has since been replaced by 13 generic versions. It is commonly prescribed to alleviate symptoms linked to upper gastrointestinal motility disorders, including diabetic gastroparesis, gastroesophageal reflux, and nausea and vomiting related to treatment for Parkinson's disease and cancer. In March 2012, Health Canada issued a warning about the potential for serious side effects associated with domperidone, such as abnormal heart rhythms and sudden cardiac death, following evidence from two studies.

Domperidone's elimination process is complex: two-thirds of the unchanged drug is excreted in feces and one-third in urine. In patients with reduced eGFR, the elimination of half-life of domperidone extends from 7 to 20 hours, prompting some prescribing guidelines to recommend a lower daily dose for those with impaired renal function. Current product monographs recommended a dose reduction for domperidone in patients with eGFR <30 mL/min/1.73 m², recommending 10 mg once or twice daily. This recommendation is based on domperidone's large volume of distribution, which means it is unlikely to be significantly removed by dialysis. Similar dosing is advised for patients on intermittent hemodialysis or peritoneal dialysis. Despite these recommendations, domperidone is still prescribed at doses over 30 mg/day, which exceeds the recommended dose for older adults with CKD in Canada.

Older adults, who are often underrepresented in clinical trials, are at increased risk for adverse drug reactions due to age-related declines in kidney function and the lack of clear prescribing dosing recommendations for patients with reduced kidney function. Population-based drug safety studies tend to focus on a single medication or a limited number of outcomes, potentially overlooking significant safety signals that could be relevant for these vulnerable patients. To address this, the investigators have developed a high-throughput computing approach to identify these signals more efficiently. This approach confirmed prior safety signals, such as the increased 30-day risk of encephalopathy with baclofen use in older patients with CKD, particularly at higher doses (≥20 mg/day) compared to lower doses (<20 mg/day) and identified new ones that warrant further investigation in another jurisdiction. Notably, preliminary findings revealed that new users of domperidone have a higher 30-day relative risk of emergency room visits, hospitalizations, and mortality compared to non-users.

To validate these findings, the investigators will conduct a population-based, new-user cohort study among patients with advanced kidney disease (eGFR <45) using linked administrative healthcare databases in Ontario, Canada, from 2008 to 2024. Additionally, the investigators will replicate this analysis using linked administrative healthcare databases in Alberta.

*Research location*

This study will utilize data from linked provincial administrative healthcare databases in Ontario and Alberta. Data for Ontario residents will be sourced from Ontario's linked administrative healthcare databases, housed and managed by ICES (ices.on.ca). The databases offer secure, encrypted data at the individual level for Ontario residents, all of whom have universal access to hospital and physician services under a government-funded, single-payer healthcare system. The use of data in this study is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a research ethics board.

The Ontario administrative datasets, which include the Canadian Institute for Health Information Discharge Abstract Database (CIHI-DAD), Ontario Drug Benefit Database (ODB), ICES Physician Database, Ontario Health Insurance Plan (OHIP) Database, National Ambulatory Care Reporting System (NACRS), Ontario Laboratories Information System (OLIS), Ontario Mental Health Reporting System (OMHRS), and the Registered Persons Database (RPDB), which are linked using unique encoded identifiers and analyzed at ICES. Trained personnel code hospital admissions and diagnoses using the 10th Revision of the International Classification of Diseases (ICD-10), relying solely on physician-documented diagnoses in patients' medical charts, without reviewing or interpreting symptoms or test results. The information required for analyzing the primary outcomes is available across specific databases within the ICES system: data on all-cause hospitalizations are available in CIHI-DAD, emergency visits in NACRS, and mortality in RPDB.

*Data Access in Alberta*

Data for each study in Alberta will be accessed in one of two ways, under the guidance of a Nephrologist and Professor of Medicine and Community Health Sciences at the University of Calgary.

1. Through the Alberta Kidney Disease Network (AKDN), Nephrologist in Alberta invited Dr. Garg to participate in prior drug safety studies that used this data source to generate new information on kidney diseases. This dataset ends in ~ 2021.
2. Through the Alberta SPOR SUPPORT Unit. Dr. Garg uses this approach with an active CIHR-funded published protocol.

As a recommended research practice, the investigators publicly document the study description, design, and statistical analysis plan on clinicaltrials.gov before analyzing the study outcomes.

*Statistical analysis plan*

Software: All statistical analyses will be conducted using SAS software version 9.4 (SAS Institute, Cary, NC).

Descriptive Statistics: Categorical variables will be reported as frequencies and proportions, while continuous variables will be presented as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate. Differences in baseline characteristics between the high-dose and low-dose groups will be examined using standardized differences, with differences ≥10% considered meaningful.

As described, the investigators will use the inverse probability of treatment weighting on the propensity score to balance baseline characteristics between the high-dose and low-dose groups.

Balancing comparator group: Inverse probability of treatment weighting on the propensity score will be used to balance characteristics between high dose (i.e., domperidone ≥30 mg/d) and low dose (i.e., domperidone <30 mg/d) groups based on their baseline characteristics, including known indicators for domperidone use. The investigators will conduct multivariable logistic regression analyses to generate propensity scores using all baseline characteristics. Patients in the low dose group will be assigned weights based on the average treatment effect for the treated, calculated as (propensity score / [1 - propensity score]). In contrast, patients in the high dose group will receive a weight of 1. This method will produce a weighted pseudo-sample of patients in the referent group (i.e., low-dose: domperidone <30 mg/day) with a similar distribution of measured characteristics as the high-dose (domperidone ≥30 mg/d) group. Baseline characteristics between groups will be compared using standardized differences in unweighted and weighted samples, with differences exceeding 10% to be considered meaningful.

Regression analysis: To evaluate the primary outcome composite measure of all-cause hospitalization or all-cause emergency department visits, or all-cause mortality- the investigators will apply a modified Poisson regression analysis to estimate the weighted risk ratio (RR) with 95% confidence intervals (CIs) and a binomial regression to estimate the weighted risk difference (RD) with 95% CIs.

Additional analysis: The investigators will conduct five additional analyses.

1. The investigators will conduct a pre-specified subgroup analysis of the primary outcome stratified by pre-2020 (which overlaps with high-throughput computing) (January 1, 2008, to March 01, 2020) and post-2020 (which does not overlap with high-throughput computing) (April 01, 2020, to September 30, 2024). Alberta data will be combined with Ontario data for the subgroup analyses.
2. The investigators will analyze the primary outcome stratified by kidney function (CKD stage using serum creatinine measurements) in patients with eGFR below 30 mL/min/1.73 m², 30-<45 mL/min/1.73 m².
3. For each cohort, the investigators will compute the hazard ratio for all outcomes within 30 days, illustrating the effect of the intervention on each outcome over time. Although the difference between hazard ratios and relative risks may be minimal over a short follow-up period, the hazard ratio offers additional insight by accounting for time-to-event analysis.
4. The investigators will conduct an analysis using a negative control exposure, the investigators will repeat the regression analyses for the initial signals, assessing the risk ratios (RRs) and risk differences (RDs) for 30-day outcomes, beginning 90 days prior to cohort entry (i.e., 90 days before the prescription start date).
5. The investigators will perform E-value analyses to determine the minimum association strength an unmeasured confounder would need with the prescription drug and the outcome of interest (while adjusting for measured covariates) to eliminate the observed association.

*Combining Outcome Results from Ontario and Alberta*

The investigators will implement one of two approaches described below to combine outcome results from Alberta and Ontario, with a preference for privacy-preserving methods, while maintaining data privacy and regulatory compliance.

1. Privacy-preserving methods: The investigators plan to use a privacy-preserving Cox-based approach for estimating risk ratios for multisite studies where individual-level data cannot be shared due to privacy constraints. The proposed method requires only a single transfer of summary-level outputs from each province to the research team. It produces results identical to those from a corresponding modified Poisson regression with combined individual-level data. The method was developed by adapting the risk-set table approach for survival outcomes, assuming stratified province-specific baseline risks, and allowing for confounding mitigation strategies such as propensity score matching or weighting to be done individually in each province. Each province will independently calculate these summary tables using their individual-level data. The summary-level risk-set tables generated in Alberta will be shared in a single data transfer to the coordinating site's analyst where they will be used to estimate the combined risk ratios and 95% confidence intervals. This will enable a robust and consistent analysis while maintaining data privacy and adhering to regulatory compliance. To comply with privacy regulations for minimizing the chance of identification of any individual, in all manuscripts, numbers of individuals are suppressed in the case of 5 or fewer participants (reported as ≤5). All team members will sign any required data confidentiality and data use agreements.

   The Alberta SPOR SUPPORT Unit recently approved this approach in a published protocol that combines Alberta and Ontario data.
2. Meta-analytic techniques: The investigators will combine risk ratios and risk differences across regions, following the methodology employed in our previous work. The investigators will first examine region-level statistical heterogeneity using the I² statistic (where an I² >50% would indicate substantial variability across regions). If substantial heterogeneity is found, the investigators will present the results of each region separately. Without substantial heterogeneity, the investigators will use meta-analytic techniques to combine the results across regions using a random effects model. Summary estimates and corresponding 95% CIs will be reported within the <45 eGFR category using appropriate methods.

ELIGIBILITY:
Inclusion Criteria:

Older adults aged 66 years or older who filled a new oral prescription for domperidone at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 1, 2008, to September 30, 2024. The investigators will exclude individuals undergoing dialysis or those who have received a kidney transplant. The age criterion is set to guarantee that individuals in this population had at least one year of prior prescription drug coverage. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once.

Exclusion Criteria:

1. Data cleaning exclusions (e.g., missing or invalid age or sex, OHIP ineligible on index date, death on or before the index date, non-Ontario residents). The investigators anticipate that very few records will be excluded due to data cleaning.
2. The investigators will exclude patients with unusual daily doses of less than 10 mg/day or >40 mg/day for domperidone. The recommended maximum daily dose for domperidone is 10 mg three times daily (30 mg/day). Some patients may require doses up to 4 times daily.
3. To ensure that patients are new domperidone users, the investigators will exclude those with any evidence of domperidone use in the 180 days before the index date.
4. Patients with more than one eligible domperidone prescription on the index date will be excluded, as this complicates the ability to ascertain the prescribed dose accurately.
5. The investigators will exclude patients with a prescription for any other prokinetic drugs and non-oral study drugs in the previous 180 days (including index date) (Note: - Gastrointestinal drugs (Cisapride, Metoclopramide, Domperidone, Prucalopride, Linaclotide)).
6. Patients with a history of kidney failure (receipt of maintenance dialysis or a kidney transplant before cohort entry).
7. The investigators will exclude patients discharged from a hospital or emergency department within the two days preceding the index date. In Ontario, when patients initiate a domperidone prescription during a hospital admission, their outpatient prescription is typically dispensed on the day they are discharged or the following day.
8. Patients with no serum creatinine measurement in the seven days prior to the year before the index date will be excluded. Patients with unstable baseline kidney function (i.e., if the most recent prior serum creatinine test was an inpatient test [ER or hospitalization] and if the corresponding eGFR differed from the most recent outpatient test by 10 mL/min/1.73 m2 or more). Previously been demonstrated that outpatient serum creatinine measurements in the province, conducted on a single occasion, indicate stable values.
9. The investigators will exclude patients with eGFR ≥45 mL/min/1.73 m² - to restrict to patients with low kidney function only.
10. If more than one eligible prescription is available, restrict it to the first. The date of this prescription will be the index date.

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults aged 66 years or older with advanced CKD who filled at least one outpatient prescription for oral domperidone between 2008 and 2024 in Ontario, and Alberta
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with a composite outcome of all-cause hospitalization or all-cause emergency visits, or all-cause mortality | Exposed cohort to domperidone (high dose (≥30 mg/d) versus low dose (<30 mg/d)) will enter the cohort between January 1, 2008, and September 30, 2024, and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  All-cause hospitalization, all-cause emergency visits, and all-cause mortality will be combined into a composite measure. Only the first hospitalization and first emergency department visit occurring after the cohort entry date will be considered.

SECONDARY OUTCOMES:
Number of participants with all-cause hospitalization | Exposed cohort to domperidone (high dose (≥30 mg/d) versus low dose (<30 mg/d)) will enter the cohort between January 1, 2008, and September 30, 2024, and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  Each component of the primary composite outcome (all-cause hospitalization, all-cause emergency department visits, and all-cause mortality) will also be presented individually as secondary outcomes. Only the first hospitalization after the cohort entry date will be considered.
Number of participants with all-cause emergency department visits | Exposed cohort to domperidone (high dose (≥30 mg/d) versus low dose (<30 mg/d)) will enter the cohort between January 1, 2008, and September 30, 2024, and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  Each component of the primary composite outcome (all-cause hospitalization, all-cause emergency department visits, and all-cause mortality) will also be presented individually as secondary outcomes. Only the first emergency department visit after the cohort entry date will be considered.
Number of participants with all-cause mortality | Exposed cohort to domperidone (high dose (≥30 mg/d) versus low dose (<30 mg/d)) will enter the cohort between January 1, 2008, and September 30, 2024, and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  Each component of the primary composite outcome (all-cause hospitalization, all-cause emergency department visits, and all-cause mortality) will also be presented individually as secondary outcomes.

OTHER OUTCOMES:
30-day hospital encounter with composite outcome of Atrial Fibrillation/flutter or ventricular arrhythmia or other arrhythmia | Exposed cohort to domperidone (high dose (≥30 mg/d) versus low dose (<30 mg/d)) will enter the cohort between January 1, 2008, and September 30, 2024, and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30- day hospital encounter (hospital admission or emergency visit) composite of Atrial fibrillation/flutter, ventricular arrhythmia/sudden cardiac death, and other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator)
30-day hospital encounter with composite outcome of delirium or falls or encephalopathy, or CT scan of the head | Exposed cohort to domperidone (high dose (≥30 mg/d) versus low dose (<30 mg/d)) will enter the cohort between January 1, 2008, and September 30, 2024, and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30- day hospital encounter (hospital admission or emergency visit) with composite outcome of delirium, falls, encephalopathy, CT scan of the head.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Higgins JP, Thompson SG, Deeks JJ, Altman DG. Measuring inconsistency in meta-analyses. BMJ. 2003 Sep 6;327(7414):557-60. doi: 10.1136/bmj.327.7414.557. PMID 12958120
- [Background] Jun M, Scaria A, Andrade J, Badve SV, Birks P, Bota SE, Campain A, Djurdjev O, Garg AX, Ha J, Harel Z, Hemmelgarn B, Hockham C, James MT, Jardine MJ, Levin A, McArthur E, Ravani P, Shao S, Sood MM, Tan Z, Tangri N, Whitlock R, Gallagher M. Kidney function and the comparative effectiveness and safety of direct oral anticoagulants vs. warfarin in adults with atrial fibrillation: a multicenter observational study. Eur Heart J Qual Care Clin Outcomes. 2023 Sep 12;9(6):621-631. doi: 10.1093/ehjqcco/qcac069. PMID 36302143
- [Background] Tangri N, Grams ME, Levey AS, Coresh J, Appel LJ, Astor BC, Chodick G, Collins AJ, Djurdjev O, Elley CR, Evans M, Garg AX, Hallan SI, Inker LA, Ito S, Jee SH, Kovesdy CP, Kronenberg F, Heerspink HJ, Marks A, Nadkarni GN, Navaneethan SD, Nelson RG, Titze S, Sarnak MJ, Stengel B, Woodward M, Iseki K; CKD Prognosis Consortium. Multinational Assessment of Accuracy of Equations for Predicting Risk of Kidney Failure: A Meta-analysis. JAMA. 2016 Jan 12;315(2):164-74. doi: 10.1001/jama.2015.18202. PMID 26757465
- [Background] Ha JT, Scaria A, Andrade J, Badve SV, Birks P, Bota SE, Campain A, Djurdjev O, Garg AX, Harel Z, Hemmelgarn B, Hockham C, James MT, Jardine MJ, Lam D, Levin A, McArthur E, Ravani P, Shao S, Sood MM, Tan Z, Tangri N, Whitlock R, Gallagher M, Jun M. Safety and Effectiveness of Rivaroxaban Versus Warfarin Across GFR Levels in Atrial Fibrillation: A Population-Based Study in Australia and Canada. Kidney Med. 2023 May 16;5(7):100675. doi: 10.1016/j.xkme.2023.100675. eCollection 2023 Jul. PMID 37492112
- [Background] Parikh RV, Nash DM, Brimble KS, Markle-Reid M, Tan TC, McArthur E, Khoshniat-Rad F, Sood MM, Zheng S, Pravoverov L, Nesrallah GE, Garg AX, Go AS. Kidney Function and Potassium Monitoring After Initiation of Renin-Angiotensin-Aldosterone System Blockade Therapy and Outcomes in 2 North American Populations. Circ Cardiovasc Qual Outcomes. 2020 Sep;13(9):e006415. doi: 10.1161/CIRCOUTCOMES.119.006415. Epub 2020 Sep 2. PMID 32873054
- [Background] Shu D, Yoshida K, Fireman BH, Toh S. Inverse probability weighted Cox model in multi-site studies without sharing individual-level data. Stat Methods Med Res. 2020 Jun;29(6):1668-1681. doi: 10.1177/0962280219869742. Epub 2019 Aug 26. PMID 31448681
- [Background] Shu D, Zou G, Hou L, Petrone AB, Maro JC, Fireman BH, Toh S, Connolly JG. A simple Cox approach to estimating risk ratios without sharing individual-level data in multisite studies. Am J Epidemiol. 2025 Jan 8;194(1):226-232. doi: 10.1093/aje/kwae188. PMID 38973755
- [Background] Haneuse S, VanderWeele TJ, Arterburn D. Using the E-Value to Assess the Potential Effect of Unmeasured Confounding in Observational Studies. JAMA. 2019 Feb 12;321(6):602-603. doi: 10.1001/jama.2018.21554. No abstract available. PMID 30676631
- [Background] Lipsitch M, Tchetgen Tchetgen E, Cohen T. Negative controls: a tool for detecting confounding and bias in observational studies. Epidemiology. 2010 May;21(3):383-8. doi: 10.1097/EDE.0b013e3181d61eeb. PMID 20335814
- [Background] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Background] Austin PC. Variance estimation when using inverse probability of treatment weighting (IPTW) with survival analysis. Stat Med. 2016 Dec 30;35(30):5642-5655. doi: 10.1002/sim.7084. Epub 2016 Aug 22. PMID 27549016
- [Background] Austin PC. An Introduction to Propensity Score Methods for Reducing the Effects of Confounding in Observational Studies. Multivariate Behav Res. 2011 May;46(3):399-424. doi: 10.1080/00273171.2011.568786. Epub 2011 Jun 8. PMID 21818162
- [Background] Brookhart MA, Wyss R, Layton JB, Sturmer T. Propensity score methods for confounding control in nonexperimental research. Circ Cardiovasc Qual Outcomes. 2013 Sep 1;6(5):604-11. doi: 10.1161/CIRCOUTCOMES.113.000359. Epub 2013 Sep 10. No abstract available. PMID 24021692
- [Background] Sato T, Matsuyama Y. Marginal structural models as a tool for standardization. Epidemiology. 2003 Nov;14(6):680-6. doi: 10.1097/01.EDE.0000081989.82616.7d. PMID 14569183
- [Background] Austin PC, Stuart EA. Moving towards best practice when using inverse probability of treatment weighting (IPTW) using the propensity score to estimate causal treatment effects in observational studies. Stat Med. 2015 Dec 10;34(28):3661-79. doi: 10.1002/sim.6607. Epub 2015 Aug 3. PMID 26238958
- [Background] Bathini L, Jeyakumar N, Sontrop J, McArthur E, Kang Y, Luo B, Bello A, Collister D, Ahmed S, Kaul P, Youngson E, Braam B, Melamed N, Hladunewich M, Garg AX. Impact of Baseline Kidney Function on the Rate of Progressive Kidney Disease After Pregnancy: A Population-Based Cohort Study Research Protocol. Can J Kidney Health Dis. 2025 Feb 28;12:20543581251318836. doi: 10.1177/20543581251318836. eCollection 2025. PMID 40027936
- [Background] Jeong R, Quinn RR, Lentine KL, Lloyd A, Ravani P, Hemmelgarn B, Braam B, Garg AX, Wen K, Wong-Chan A, Gourishankar S, Lam NN. Outcomes Following Macrolide Use in Kidney Transplant Recipients. Can J Kidney Health Dis. 2019 Feb 21;6:2054358119830706. doi: 10.1177/2054358119830706. eCollection 2019. PMID 30815270
- [Background] Muanda FT, Weir MA, Bathini L, Blake PG, Chauvin K, Dixon SN, McArthur E, Sontrop JM, Moist L, Garg AX. Association of Baclofen With Encephalopathy in Patients With Chronic Kidney Disease. JAMA. 2019 Nov 26;322(20):1987-1995. doi: 10.1001/jama.2019.17725. PMID 31705755
- [Background] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562
- [Background] Rojas-Fernandez C, Stephenson AL, Fischer HD, Wang X, Mestre T, Hutson JR, Pondal M, Lee DS, Rochon PA, Marras C. Current use of domperidone and co-prescribing of medications that increase its arrhythmogenic potential among older adults: a population-based cohort study in Ontario, Canada. Drugs Aging. 2014 Nov;31(11):805-13. doi: 10.1007/s40266-014-0215-z. PMID 25227452
- [Background] Reddymasu SC, Soykan I, McCallum RW. Domperidone: review of pharmacology and clinical applications in gastroenterology. Am J Gastroenterol. 2007 Sep;102(9):2036-45. doi: 10.1111/j.1572-0241.2007.01255.x. Epub 2007 May 3. PMID 17488253
- [Background] Expert opinion. Senior Renal Editorial Team: Bruce Mueller, PharmD, FCCP, FASN, FNKF; Jason A. Roberts, PhD, BPharm (Hons), B App Sc, FSHP, FISAC; Michael Heung, MD, MS.
- [Background] Johannes CB, Varas-Lorenzo C, McQuay LJ, Midkiff KD, Fife D. Risk of serious ventricular arrhythmia and sudden cardiac death in a cohort of users of domperidone: a nested case-control study. Pharmacoepidemiol Drug Saf. 2010 Sep;19(9):881-8. doi: 10.1002/pds.2016. PMID 20652862
- [Background] van Noord C, Dieleman JP, van Herpen G, Verhamme K, Sturkenboom MC. Domperidone and ventricular arrhythmia or sudden cardiac death: a population-based case-control study in the Netherlands. Drug Saf. 2010 Nov 1;33(11):1003-14. doi: 10.2165/11536840-000000000-00000. PMID 20925438
- [Background] Drolet B, Rousseau G, Daleau P, Cardinal R, Turgeon J. Domperidone should not be considered a no-risk alternative to cisapride in the treatment of gastrointestinal motility disorders. Circulation. 2000 Oct 17;102(16):1883-5. doi: 10.1161/01.cir.102.16.1883. PMID 11034933
- [Background] Barone JA. Domperidone: a peripherally acting dopamine2-receptor antagonist. Ann Pharmacother. 1999 Apr;33(4):429-40. doi: 10.1345/aph.18003. PMID 10332535
- [Background] Rossi M, Giorgi G. Domperidone and long QT syndrome. Curr Drug Saf. 2010 Jul 2;5(3):257-62. doi: 10.2174/157488610791698334. PMID 20394569
- [Background] Doggrell SA, Hancox JC. Cardiac safety concerns for domperidone, an antiemetic and prokinetic, and galactogogue medicine. Expert Opin Drug Saf. 2014 Jan;13(1):131-8. doi: 10.1517/14740338.2014.851193. Epub 2013 Oct 23. PMID 24147629
- See also: Government of Canada. Summary Safety Review - DOMPERIDONE - Serious abnormal heart rhythms and sudden death (cardiac arrest) — https://dhpp.hpfb-dgpsa.ca/review-documents/resource/SSR00039
- See also: Domperidone: Drug information - UpToDate — https://online-lexi-com.proxy.lib.uwaterloo.ca/lco/action/doc/retrieve/docid/patch_f/6782?cesid=8oJ5rWaJfSj&searchUrl=%2Flco%2Faction%2Fsearch%3Fq%3Ddomperidone%26t%3Dname%26acs%3Dfalse%26acq%3Ddomperidone
- See also: Domperidone (Product Monograph) — https://pdf.hres.ca/dpd_pm/00070468.PDF
- See also: CPS [Internet]. Ottawa (ON): Canadian Pharmacists Association; c2017 [updated 2017, November 01]. Domperidone [product monograph] — https://cps-pharmacists-ca.proxy.lib.uwaterloo.ca/search
- See also: ICES. ICES data [Internet] — https://www.ices.on.ca/